CLINICAL TRIAL: NCT06314776
Title: Whole-Body Vibration Therapy in the Gait of Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María del Mar Sánchez Joya, Associate Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEURO24
Record Dates: First submitted 2024-03-09; First posted 2024-03-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy; Neurologic Disorder; Gait Disorders in Children; Hemiplegia
Keywords: Cerebral Palsy; Whole-Body Vibration
MeSH Terms: conditions — Cerebral Palsy; Nervous System Diseases; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Usual physiotherapy (Active Comparator): Pre-intervention (GMFM, Test 10M, Test Time Up and Go)
  Interventions: Other: Pre-Usual physiotherapy
- Usual physiotherapy without Whole-Body Vibration (Active Comparator): Two days a week of physical therapy (mobilizations, manual therapy, stretching, respiratory techniques)
  Interventions: Other: Usual physiotherapy without Whole-Body Vibration
- Post-Usual physiotherapy (Active Comparator): Post-intervention (GMFM, Test 10M, Test Time Up and Go)
  Interventions: Other: Post-Usual physiotherapy

INTERVENTIONS:
Other: Usual physiotherapy without Whole-Body Vibration — Manual Therapy, passive and active mobilizations, stretching, respiratory techniques
  Arms: Usual physiotherapy without Whole-Body Vibration
Other: Pre-Usual physiotherapy — (GMFM, Test 10M, Test Time Up and Go)
  Arms: Pre-Usual physiotherapy
Other: Post-Usual physiotherapy — (GMFM, Test 10M, Test Time Up and Go)
  Arms: Post-Usual physiotherapy

SUMMARY:
Observation of the effect of vibration therapy on the gait of children with cerebral palsy and the analysis of their functional evolution

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neurological developmental disorder: Cerebral Palsy. (According to DSM-V)
* Age between 2 to 11 years.
* GMFCS I and II.
* Assessed and/or intervened in or from centers, institutions, etc. who collaborate with the University of Almería or participate in them. Specifically from the "Interactúa" Child Development and Early Care Center.
* The subject, father/mother/legal guardian of each subject, prior to inclusion in the study, must have signed the informed consent for the participation of himself or his/her child in it, leaving a record that it could be abandoned if at any time they deem it appropriate and without having to justify it.

Exclusion Criteria:

* Diagnosis of Epilepsy.
* Serious blood circulation problems.
* Recent operations.
* Prosthetics.
* Start of another type of therapy different from the current one.
* Not having indication for Physiotherapy.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Test Time Up and Go | One Month
  The time it takes children to walk 3 metres, getting up from a standard chair walking to a cone and back and sitting back down is measured. The result of this scale is the time that the children take to do this, if the time decrease after the time of intervention that means the children improve their physical condition.
Timed 10-Meter Walk Test | One Month
  The time traveled in seconds over a distance is measured, from the 2 meter mark to meter 8 is taken into consideration, three attempts are made by each participant. The result of this scale is the time that the children take to do this, if the time decrease after the time of intervention that means the children improve their physical condition.
Gross Motor Function Measure | One Month
  This scale consists of an 88 items test to assess gross motor function, as higher score have the children better physical condition.

CONTACTS AND LOCATIONS:
Locations (1):
- María del Mar Sánchez-Joya, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: SAP
Time Frame: Data will become available for one year once the study is finished
Access Criteria: Reasonable request to reproduce the intervention performed on this study